CLINICAL TRIAL: NCT05294653
Title: Risk of Atherosclerotic Cardiovascular Disease in Childhood and Teen-age Onset Diabetes
Brief Title: Atherosclerotic Cardiovascular Risk in Childhood and Teen-age Onset Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Weiqiong Gu, Risk of Atherosclerotic Cardiovascular Disease in Childhood and Teen-age Onset Diabetes, Shanghai Jiao Tong University School of Medicine
Other Study IDs: youngascvd
Record Dates: First submitted 2022-02-25; First posted 2022-03-24 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Atherosclerotic Cardiovascular Disease; Childhood Diabetes Mellitus; Juvenile Diabetes
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 1 Diabetes: Classified according to American Diabetes Association [ADA] 2021 guidelines
- Type 2 Diabetes: Classified according to American Diabetes Association [ADA] 2021 guidelines

SUMMARY:
For children and adolescents with diabetes, the pathological process of atherosclerotic cardiovascular disease(ASCVD) can exist in early childhood and progress rapidly to subclinical ASCVD. This study intends to explore the models for the prediction of ASCVD risk in childhood and teen-age onset diabetes with different types.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease (ASCVD) is the main cause of death in patients with diabetes. Currently recognized ASCVD risk assessment models are limited to adults with diabetes, but for children and adolescents with diabetes, the pathological process of ASCVD can exist in early childhood and progress rapidly to subclinical ASCVD.

To sum up, this study intends to evaluate the high risk rate of ASCVD calculated by the traditional QRISK3 model and its correlation with the occurrence of subclinical ASCVD events through long-term follow-up of the natural history of diabetes onset in children and adolescents, and to explore the models for the prediction of ASCVD risk in childhood and teen-age onset diabetes with different types. This study aims to help block the pathological process of ASCVD in early duration, thereby reducing the occurrence of ASCVD in childhood and teen-age onset diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 1 diabetes or type 2 diabetes
2. Age of onset: <18y
3. Enrollment age: ≥18y
4. Gender: male or female
5. Diabetes duration ≥ 5 years

Exclusion Criteria:

1. Specific types of diabetes
2. Clinical diagnosis of diabetes is unknown, and it belongs to untyped diabetes
3. Pregnancy or lactation
4. Received glucocorticoids, immunosuppressants, non-glycemic biological agents, and cytotoxic drugs in the past 3 months; non-steroidal pain relievers or antibiotics used for more than 1 week continuously
5. Onset of acute complications of diabetes in the past 3 months
6. Major trauma and surgery history in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Random
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Atherosclerotic Cardiovascular Disease(ASCVD) high risk rating | 5 years
  Risk value calculated by QRISK3 model >10% (The QRISK®3-2018 risk calculator https://qrisk.org/three)

SECONDARY OUTCOMES:
Occurrence of subclinical ASCVD(carotid plaque) | 5 years
  Carotid plaque(IMT>1.5mm)
Occurrence of subclinical ASCVD(carotid intima-media thickness) | 5 years
  Carotid intima-media thickness(CIMT)≥0.9mm
Occurrence of subclinical ASCVD(pulse wave velocity) | 5 years
  Pulse wave velocity(PWV)>6.8m/s
Occurrence of subclinical ASCVD(coronary artery calcium) | 5 years
  Coronary artery calcium(CAC) score>0 (CAC:assessed only when subclinical ASCVD events confirmed by IMT, CIMT, PWV)

OTHER OUTCOMES:
Glycemic control(glycated hemoglobin) | 5 years
  To study glycemic control by comparing glycated hemoglobin(HbA1c)
Glycemic control(free blood glucose) | 5 years
  To study glycemic control by comparing free blood glucose(FBG)
Glycemic control(postprandial blood glucose) | 5 years
  To study glycemic control by comparing postprandial blood glucose(PBG) with mixed meal tolerance test (MMTT)
Glycemic control(severe hypoglycemia events) | 5 years
  Severe hypoglycemia events in the past six months
Islet function(fasting C peptide) | 5 years
  To study the residual β-cell function by using fasting C peptide(FCP)
Islet function(2-hour post-meal stimulated C peptide) | 5 years
  To study the residual β-cell function by using 2-hour post-meal stimulated C peptide (PCP) with MMTT
Islet function(pancreatic enhanced MR) | 5 years
  Volume of the pancreas(ml) calculated by pancreatic enhanced MR
Daily insulin dosage | 5 years
  To study the insulin requirement by using daily insulin dosage per body weight (DID IU/kg.d)
Frequency of daily moderate to high-intensity aerobic exercise | 5 years
  To assess the influence of exercise by measuring the frequency of daily moderate to high-intensity aerobic exercise (<60min, ≥60min) [pulse=(220-age)*(60-75%)]
Occurrence of diabetic nephropathy | 5 years
  Urine microalbumin (MA)/creatinine (Cr) ratio
Concentration of cardiac troponin T | 5 years
  To assess the myocardial function by cardiac troponin T(cTnI)
Level of high-sensitivity C-reactive protein | 5 years
  To assess the extent of inflammation by high-sensitivity C-reactive protein (hs-CRP)
Occurrence of diabetic retinopathy | 5 years
  Retinal photography
Level of cardiac function | 5 years
  Echocardiography
Occurrence of diabetic neuropathy | 5 years
  Electrophysiological testing
Level of thyroid hormones | 5 years
  To assess the occurrence of thyroiditis by thyroid function including triiodothyronine, tetraiodothyronine, thyroid stimulating hormone and thyroid autoantibodies
Level of free cortisol rhythm | 5 years
  To assess the function of adrenal gland by measuring the level of free cortisol rhythm
Occurrence of rheumatic diseases | 5 years
  Rheumatic antibody

CONTACTS AND LOCATIONS:
Overall Officials: Weiqiong Gu, PhD, Principal Investigator — Department of Endocrinology and Metabolic Diseases, Ruijin Hospital, Shanghai Jiao-Tong University
Locations (1):
- Department of Endocrinology and Metabolic Diseases, Ruijin Hospital, Shanghai Jiao-Tong University, Shanghai, China